CLINICAL TRIAL: NCT05282888
Title: ERYthrocyte Morphology Using Flow Imaging on ImageSTREAM Cytometer
Acronym: ERYSTREAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0087
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Red Blood Cells; Schistocytes; Artificial Intelligence
Keywords: Red blood cells; schistocytes; flow imaging; artificial intelligence
MeSH Terms: conditions — Sickle Cell Trait | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood withdrawal in order to study red blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample — in order to develop a diagnostic assay using an innovative technology by imaging flow cytometry to identify red blood cell morphological anomalies in the diagnosis flowchart of anemia.

SUMMARY:
Erythrocyte morphology analysis is a key step in the diagnosis flowchart of anemia. It is performed on a peripheral blood smear after May Grümwald Giemsa staining. In the context of hemolytic anemias for example, it allows the recognition of therapeutic emergencies such as sickle cell disease crisis, malaria-induced hemolysis and thrombotic microangiopathy, the latter being characterized by the presence of schistocytes and justifying an immediate clinical care. However, cytological analysis of erythrocyte morphology requires pre-analytical interventions (smear spreading + staining), the quality of which determines the accuracy of the result. Moreover, it requires a good cytological expertise and may be sometimes subjective. For several years, alternative methods for erythrocyte morphology evaluation have been developed, based on automated hematology machines or automated microscopy. Nevertheless, none of them has yet proven itself in comparison with cytology, especially in the diagnosis of thrombotic microangiopathies. By combining the advantages of flow cytometry and microscopy, flow imaging appears to be a promising technology for the diagnosis of anemias: it does not require any pre-analytical intervention, does not require any spreading and analyzes a large number of events. Moreover, it can be coupled with artificial intelligence via the generation of an apprenticeship by the constitution of a large image data base, which then allows the recognition of the different red blood cells morphologies without human eyes. The objective of this study is to build a data base containing the main red blood cell morphologies relevant in anemia, and to validate it through a comparison in anemic patients of erythrocyte morphological assessment either directly on whole blood by flow imaging or routinely by cytological analysis of peripheral blood smear after by a trained operator.

ELIGIBILITY:
Inclusion Criteria:

* Any patient for whom a blood test including a cytological evaluation of RBC morphology is performed in the routine laboratory of CHU Amiens

Exclusion Criteria:

* patients who have opposed the use of their personal data for research work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient for whom a blood test including a cytological evaluation of RBC morphology is performed in the routine laboratory of CHU Amiens
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Concordance between classical cytological erythrocyte analysis and ImageStream flow imaging erythrocyte analysis | 6 months
  The investigators will characterize by flow imaging the normal and pathological erythrocyte morphologies by creating a bank of images representative of the main red blood cell abnormalities observed during anemias. The images will be classified manually by the investigators in order to create a morphological data base allowing apprenticeship via artificial intelligence. Once the database will be created, the investigators will validate it prospectively by comparison between classical cytological analysis and flow imaging on samples for which a blood test will be prescribed for anemia.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No